CLINICAL TRIAL: NCT00810641
Title: Randomized Multicenter Study of Treatment of Horizontal Canal Benign Paroxysmal Positional Vertigo
Brief Title: Treatment of Apogeotropic Horizontal Canal Benign Paroxysmal Positional Vertigo
Acronym: BPPV-HC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chonbuk National University (Other)
Collaborators: Seoul National University Bundang Hospital (Other)
Responsible Party: KONOS, Korean neuro-ophthalmology and neuro-otology society
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KONOS
Record Dates: First submitted 2008-12-17; First posted 2008-12-18 (Estimated); Results first posted 2011-06-27 (Estimated); Last update posted 2011-06-27 (Estimated); Status verified 2011-05

CONDITIONS: HC-BPPV
Keywords: BPPV(benign paroxysmal positional vertigo); HC-BPPV(BPPV involving the horizontal semicircular canal); Nystagmus; Treatment outcome; Horizontal Canal Benign Paroxysmal Positional Vertigo
MeSH Terms: conditions — Benign Paroxysmal Positional Vertigo; Nystagmus, Pathologic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Gufoni maneuver (Active Comparator): Gufoni maneuver for apogeotropic HC-BPPV
  Interventions: Procedure: Gufoni maneuver
- Headshaking maneuver (Active Comparator): headshaking maneuver for apogeotropic HC BPPV
  Interventions: Procedure: Head-shaking maneuver
- sham maneuver (Sham Comparator): sham maneuver for apogeotropic HC BPPV
  Interventions: Procedure: sham maneuver

INTERVENTIONS:
Procedure: Gufoni maneuver — For Gufoni maneuver,16,18 the patient was quickly brought down to the side-lying position on the affected ear from the sitting position. After one minute in this position, the head of the patient was quickly turned 45O upward, so that the nose directed upward. Approximately 2 minutes later, the patient was returned to the upright position (Figure 2A).
  Arms: Gufoni maneuver
Procedure: Head-shaking maneuver — For head-shaking maneuver,15 patients were brought into a sitting position. After pitching the head forward by approximately 30O, we moved the head sideways in a sinusoidal fashion at an approximate rate of 3 Hz for 15 seconds.
  Arms: Headshaking maneuver
Procedure: sham maneuver — For the sham maneuver, patients quickly lied on the unaffected side, and returned to the sitting position after one minute.
  Arms: sham maneuver

SUMMARY:
The purpose of this study was to compare the immediate efficacies of each treatment maneuvers in treatment of apogeotropic horizontal canal benign paroxysmal positional vertigo (HC-BPPV).

DETAILED DESCRIPTION:
A randomized prospective study of patients with HC-BPPV. Patients with apogeotropic type of HC-BPPV were randomized to one of each three treatment groups at their first clinic visit. These groups included the Gufoni maneuver, head-shaking maneuver, and sham group in apogeotropic HC-BPPV. Responsiveness of treatment maneuver was determined by positioning maneuver immediately after each treatment method based on resolves of vertigo and positional nystagmus.

ELIGIBILITY:
Inclusion Criteria:

* a history of brief episodes of positional vertigo,
* direction-changing horizontal nystagmus beating toward the uppermost (apogeotropic nystagmus) or undermost (geotropic nystagmus) ear in both the lateral head turning positions,
* no spontaneous nystagmus during upright sitting position, and
* absence of identifiable central nervous system disorders that could explain the positional vertigo and nystagmus.

Exclusion Criteria:

* central positional nystagmus with identifiable CNS lesions that could explain the positional nystagmus

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2009-01; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- South Korea (2):
  - Chonbuk National University Hospital, Jeonju, Cholabuk-do
  - Seoul National University Bundang Hospital, Seongnam, Kyoungki-do

REFERENCES:
- [Derived] Kim JS, Oh SY, Lee SH, Kang JH, Kim DU, Jeong SH, Choi KD, Moon IS, Kim BK, Oh HJ, Kim HJ. Randomized clinical trial for apogeotropic horizontal canal benign paroxysmal positional vertigo. Neurology. 2012 Jan 17;78(3):159-66. doi: 10.1212/WNL.0b013e31823fcd26. Epub 2011 Dec 14. PMID 22170885

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between February 2009 and October 2009, consecutive patients with a diagnosis of apogeotropic HC-BPPV were recruited from nationwide 10 Dizziness Clinics in Korea.
Pre-assignment Details: We defined the transition as a conversion into another canal type of BPPV without intervening periods of remission. In contrast, recurrence was defined as a redevelopment of any type of BPPV after a confirmed resolution of the positioning nystagmus and vertigo.
Groups:
- Sham Maneuver: sham maneuver for apogeotropci HC BPPV
Period: Overall Study
Arm/Group | Gufoni Maneuver | Headshaking Maneuver | Sham Maneuver
Started | 52 | 54 | 51
Completed | 52 | 53 | 49
Not Completed | 0 | 1 | 2
Not completed — Withdrawal by Subject | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Gufoni Maneuver | Headshaking Maneuver | Sham Maneuver | Total
Number analyzed (Participants) | 52 | 54 | 51 | 157
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 0 | 0 | 1
  Between 18 and 65 years | 32 | 30 | 27 | 89
  >=65 years | 19 | 24 | 24 | 67
Age Continuous [Mean (Standard Deviation); unit: years] | 57.8 (13.5) | 60.5 (12.4) | 61.5 (14.9) | 59.9 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 30 | 28 | 97
  Male | 13 | 24 | 23 | 60
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 52 | 54 | 51 | 157

OUTCOME MEASURES:

1. Primary Outcome: Treatment of Apogeotropic Horizontal Canal Benign Paroxysmal Positional Vertigo: A Randomized Clinical Trial
Description: The immediate treatment response was determined by participating neurologists in each clinic without knowing the maneuver applied to each patient from 30 minutes to one hour after initial maneuver. The absence of both vertigo and nystagmus was required to determine a resolution.
Time Frame: one hour
Population: Of the 157 patients enrolled in the study, three were lost for follow-up (dropout rate, 1.9%) and 154 were finally included for analyses.
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | Gufoni Maneuver | Headshaking Maneuver | Sham Maneuver
Number analyzed (Participants) | 52 | 53 | 49
participants | 38 [2.48 to 13.78] | 33 [1.42 to 7.17] | 17 [1.78 to 9.85]

ADVERSE EVENTS:
Arm/Group | Gufoni Maneuver | Headshaking Maneuver | Sham Maneuver
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
In this study, resolution of BPPV was determined using a telephone interview during the follow-ups after one week.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No